CLINICAL TRIAL: NCT01345032
Title: The Effect of Follow up on Nutrition Intervention After Discharge in Undernourished Geriatric Patients
Brief Title: The Effect of Nutrition Follow up After Hospital Discharge in Undernourished Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Jette Lindegaard Pedersen, Clinical research nurse, Aarhus University Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 23012011
Record Dates: First submitted 2011-04-28; First posted 2011-04-29 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Under Nutrition
MeSH Terms: interventions — House Calls; Home Environment; Home Care Services

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Home visits (Experimental): Nutritional follow-up after discharge, conducted as nutritional counselling performed as in-person counselling in the participants homes
  Interventions: Other: Home visit
- Telephone consultation (Experimental): Nutritional follow-up after discharge, conducted as nutritional counselling performed as telephone consultation
  Interventions: Other: Telephone consultation
- Control (No Intervention): No follow-up after discharge

INTERVENTIONS:
Other: Home visit — Patients and their homecare helper will receive visits from a clinical dietician 1 week, 2 weeks and 4 weeks after discharge. The purpose of the visits is follow up on the individual diet plan distributed at discharge and supply dietary advice.
  Other Names: Aged 75 and over; Living alone; Receive help for home care services; Dietary advice after discharge by home visits
  Arms: Home visits
Other: Telephone consultation — Patients and their homecare helper will be contacted on telephone from a clinical dietician 1 week, 2 weeks and 4 weeks after discharge. The purpose of the telephone contact is follow up on the individual diet plan distributed at discharge and supply dietary advice.
  Other Names: Aged 75 and over; Living alone; Receive help for home care services; Dietary advice after discharge by telephone consultation
  Arms: Telephone consultation

SUMMARY:
The purpose of this study is to test two different interventions of nutrition follow up after discharge from geriatric ward in undernourished geriatric patients. The patients are randomized to a home visit arm, a telephone consultation arm, or a control arm. Patients in the home visit arm and their home care helper will get visits from a clinical dietician at one week, two weeks and four weeks after discharge, in order to follow up on the nutrition intervention. Patients in the telephone consultation arm and their home care helper will be contacted by a clinical dietician at one week, two weeks and four weeks after discharge, in order to follow up on the nutrition intervention. The control arm will not be contacted.

The primarily outcome is functional ability. Secondary outcomes are quality of life, readmission and mortality.

DETAILED DESCRIPTION:
Under nutrition among geriatric patients is a recurrent and well documented problem. Up to 55 % of the elderly are undernourished at the time of admission. Hospitalisation and acute illness are associated to loss of muscles and physical ability, complications, dependency, morbidity and mortality. Elderly who live alone are more vulnerable to nutritional problems, than elderly who live together with another person or in a nursing home. Geriatric patients, who are admitted to geriatric ward Aarhus University Hospital due to various acute somatic disorders, aged 75 and older and who are living alone with help from the home care facilities can participate in the study. According to the power calculation 150 patients must be included, 50 patients in each arm of the study. Informed consent will be obtained before inclusion and discharge from hospital. Randomization will be computerised and determine if the patient will be allocated to the "home visit" group, the "telephone consultation" group or the "control group". Patients who suffer from mental disorder (MMSE<22) or active cancer are excluded as well as patients who live together with another person or live in a nursing home. During hospitalisation the three groups will receive the same nutritional care as all patients in nutritional risk. This includes nutritional intervention during hospitalization and an individual diet plan at discharge. Patients in the home visit arm will get visits from a clinical dietician at one week, two weeks and four weeks after discharge. Patients in the telephone consultation arm will be contacted by a clinical dietician at one week, two weeks and four weeks after discharge. In both intervention groups the patients and their home care helpers will get dietary advice and follow up on their individual diet plan. The main outcome is functional ability from discharge and to 8 weeks after discharge. Secondary outcomes are quality of life, readmission at 30 and 90 days and mortality at 30 and 90 days.

ELIGIBILITY:
Inclusion Criteria:

* aged 75 and over
* undernourished according to Mini Nutritional Assessment (MNA)
* living alone in own home
* admitted and discharged from geriatric ward Aarhus, Denmark, due to various acute somatic disorders

Exclusion Criteria:

* active cancer
* mental disorder (MMSE<22)
* live together with another person
* live in a nursing home

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 208 (Actual)
Dates: Start 2011-06; Primary Completion 2014-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Functional ability. | Between discharge and 8 weeks after discharge
  Measurements: Barthel-100 Index, Cumulated Ambulation Score (CAS), handgrip strength, part of senior fitness test,fatigue test (Avlund)

SECONDARY OUTCOMES:
Quality of Life | Between discharge and 8 weeks after discharge
  Measurements: SF-36, geriatric depression score (GDS), depression list (DL)
Mortality | Between discharge and 30 after discharge
Readmission to hospital | Between discharge and 30 days after discharge
Readmission | Between discharge and 90 days after discharge
Mortality | Between discharge and 90 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jette Lindegaard Pedersen, MHSc., Principal Investigator — Aarhus University Hospital; Else Marie S. Damsgaard, Professor, Study Chair — Aarhus University Hospital; Preben Ulrich Pedersen, Ph.D., Study Chair — University of Aarhus
Locations (2):
- Denmark (2):
  - Aarhus Universityhospital, Geriatric Department, Aarhus
  - Geriatric Department, Aarhus